CLINICAL TRIAL: NCT01540318
Title: Utility of Abdominal Ultrasound in the Evaluation of Children With Blunt Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 244545; H34MC19682 (Other Grant/Funding Number: US Department of Health and Human Services); 244545 (Other: UC Davis)
Record Dates: First submitted 2012-01-31; First posted 2012-02-28 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Abdominal Injuries
Keywords: ultrasonography; Abdominal Injuries; Trauma
MeSH Terms: conditions — Abdominal Injuries; Wounds and Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal Ultrasound (Experimental): Patients in the experimental arm will receive a "Focused Assessment with Sonography for Trauma (FAST)" which includes the use of abdominal ultrasound.
  Interventions: Procedure: Abdominal Ultrasound (FAST examination)
- No Abdominal Ultrasound (No Intervention)

INTERVENTIONS:
Procedure: Abdominal Ultrasound (FAST examination) — Use of FAST abdominal ultrasound exam
  Other Names: Focused Assesment with Sonography for Trauma
  Arms: Abdominal Ultrasound

SUMMARY:
The major goal of this project is to conduct a randomized controlled trial studying an initial evaluation strategy with abdominal ultrasound versus a strategy without abdominal ultrasound for the evaluation of children with blunt abdominal trauma. The proposal's objectives are to compare the following variables in those that randomize to abdominal ultrasound versus those that do not:

1. rate of abdominal CT scanning
2. time to emergency department disposition
3. the rate of missed/delayed diagnosis of intra-abdominal injury
4. the costs.

ELIGIBILITY:
Inclusion Criteria:

* Blunt torso trauma resulting from a significant mechanism of injury

  * Motor vehicle collision: greater than 60 mph, ejection, or rollover
  * Automobile versus pedestrian/bicycle: automobile speed > 25 mph
  * Falls greater than 20 feet in height
  * Crush injury to the torso
  * Physical assault involving the abdomen
  * Decreased level of consciousness (Glasgow Coma Scale score < 15 or below age-appropriate behavior) in association with blunt torso trauma
* Blunt traumatic event with any of the following (regardless of the mechanism):

  * Extremity paralysis
  * Multiple long bone fractures (e.g., tibia and humerus fracture)
* History and physical examination suggestive of intra-abdominal injury following blunt torso trauma of any mechanism (including mechanisms of injury of less severity than mentioned above)

Exclusion Criteria:

* No concern for inter-abdominal injury or no planned evaluation for possible IAI
* Prehospital or ED age adjusted Hypotension
* Prehospital or initial ED GCS score ≤ 8
* Presence of an abdominal "seat belt sign" - continuous area of erythema/contusion completely across the lower abdomen secondary to a lap belt
* Penetrating trauma: stab or gunshot wounds
* Traumatic injury occurring > 24 hours prior to the time of presentation to the ED
* Transfer of the patient to the UCDMC ED from an outside facility with abdominal CT scan, diagnostic peritoneal lavage, or laparotomy previously performed
* Patients with known disease processes resulting in intraperitoneal fluid including liver failure and the presence of ventriculoperitoneal shunts

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 925 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of Abdominal CT Scan | One week from enrollment

SECONDARY OUTCOMES:
Total time spent in the Emergency Department | 24 hours from enrollment
Cost effectiveness | two months from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: James F Holmes, MD, MPH, Principal Investigator — UC Davis School of Medicine
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Holmes JF, Kelley KM, Wootton-Gorges SL, Utter GH, Abramson LP, Rose JS, Tancredi DJ, Kuppermann N. Effect of Abdominal Ultrasound on Clinical Care, Outcomes, and Resource Use Among Children With Blunt Torso Trauma: A Randomized Clinical Trial. JAMA. 2017 Jun 13;317(22):2290-2296. doi: 10.1001/jama.2017.6322. PMID 28609532